CLINICAL TRIAL: NCT04683939
Title: Phase I/IIa, First-in-human, Open-label, Dose Escalation Trial With Expansion Cohorts to Evaluate Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of BNT141 as a Monotherapy and in Combination With Other Anti-cancer Agents in Patients With CLDN18.2-positive Solid Tumors
Brief Title: Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy Trial of BNT141 in Patients With Unresectable or Metastatic CLDN18.2-positive Gastric, Pancreatic, Ovarian and Biliary Tract Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT141-01; 2022-001843-25 (EudraCT Number)
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma; Pancreatic Cancer; Biliary Tract Cancer; Cholangiocarcinoma; Metastatic Cancer
Keywords: CLDN18.2-positive solid tumors; Gastric cancer; Gastric adenocarcinoma; Gastroesophageal junction adenocarcinoma; Esophageal adenocarcinoma; Esophageal cancer; Pancreatic cancer; Pancreatic ductal adenocarcinoma; Biliary tract cancers; Cholangiocarcinoma; Mucinous ovarian cancers; Metastatic; Treatment; Therapy; Targeted immunotherapy; Metastatic cancer; Ribomab; CLDN18.2-positive tumors; Biomarker; Precision medicine; Precision oncology; Solid tumors; mRNA
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma Of Esophagus; Pancreatic Neoplasms; Biliary Tract Neoplasms; Cholangiocarcinoma; Neoplasm Metastasis; Esophageal Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A - BNT141 monotherapy escalation (Experimental): Administration once every three weeks (Q3W)
  Interventions: Drug: BNT141
- Part 1B - BNT141 in combination with nab-paclitaxel and gemcitabine (Experimental): BNT141 was planned to be administered Q3W. Nab-paclitaxel and gemcitabine was planned to be administered on three days of each 28-day cycle.
  Interventions: Drug: BNT141; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Part 2 - predefined expansion cohorts (Experimental): BNT141 in combination with nab-paclitaxel and gemcitabine
  Interventions: Drug: BNT141; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: BNT141 — Intravenous (IV)
Drug: Nab-paclitaxel — IV
  Arms: Part 1B - BNT141 in combination with nab-paclitaxel and gemcitabine; Part 2 - predefined expansion cohorts
Drug: Gemcitabine — IV
  Arms: Part 1B - BNT141 in combination with nab-paclitaxel and gemcitabine; Part 2 - predefined expansion cohorts

SUMMARY:
This study was planned as an open-label, multi-site, Phase I/IIa dose escalation, safety, and pharmacokinetic (PK) trial of BNT141 followed by expansion cohorts in patients with Claudin 18.2 (CLDN18.2)-positive tumors.

The sponsor decided to stop the development of BNT141 on 24 July 2023 and the study was terminated early.

DETAILED DESCRIPTION:
The study design consisted of three parts:

* Part 1A was a dose escalation of BNT141 as monotherapy in patients with advanced unresectable or metastatic CLDN18.2-positive solid tumors for which there was no available standard therapy considered to confer clinical benefit, or the patient was not a candidate for such available therapy. The dose of BNT141 was planned to be escalated until the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of BNT141 as monotherapy was defined. However, due to the early study termination, the dose of BNT141 was not fully escalated as planned per protocol (i.e., only four doses were tested, i.e., 0.15 mg/kg, 0.30 mg/kg, 0.45 mg/kg, and 0.60 mg/kg). Once the MTD was reached, up to 10 additional patients with CLDN18.2 expressing pancreatic and biliary tract cancers were planned to be enrolled at the MTD level to obtain additional data on safety, PK and pharmacodynamics (PD). Eligible tumor types were gastric cancer, gastroesophageal junction (GEJ) and esophageal adenocarcinoma, pancreatic, biliary tract (cholangiocarcinoma and gallbladder cancer), and mucinous ovarian cancers. Additionally, patients with specific tumors (including colorectal cancer, non-small-cell lung cancer, gastric subtype of endocervical adenocarcinoma) where there is scientific evidence that the CLDN18.2 could be elevated could be tested for CLDN18.2 expression.
* Part 1B was planned to be a dose escalation of BNT141 in combination with nab-paclitaxel and gemcitabine in patients with locally advanced unresectable or metastatic CLDN18.2-positive pancreatic adenocarcinoma or cholangiocarcinoma who were eligible for treatment with nab-paclitaxel and gemcitabine. Part 1B intended to define the MTD and/or RP2D of the combination. Once the MTD was reached, up to 10 additional patients with CLDN18.2-expressing pancreatic adenocarcinoma or cholangiocarcinoma were planned to be enrolled at the MTD level to obtain additional data on safety, PK and PD. The MTD of BNT141 in combination with nab-paclitaxel and gemcitabine in Part 1B was planned to not exceed the monotherapy BNT141 MTD determined in Part 1A.
* Part 2 (Expansion) was planned to consist of two predefined expansion cohorts in patients with CLDN18.2-positive solid tumors eligible for treatment with nab-paclitaxel and gemcitabine.

Part 1B and Part 2 did not proceed and no participant was enrolled in Part 1B and Part 2.

ELIGIBILITY:
Key inclusion criteria:

For all Parts:

* Metastatic or unresectable solid tumor.
* Histological or cytological documentation of a solid tumor via a pathology report.
* CLDN18.2-positive tumor sample defined as moderate-to-strong CLDN18.2 protein expression defined as intermediate (2+) to strong (3+) staining intensity in ≥ 50% of tumor cells as assessed by central testing using a CLIA-validated immunohistochemistry assay in formalin-fixed, paraffin-embedded (FFPE) neoplastic tissues. New biopsies and archival bio-samples are allowed. Bone biopsies are not allowed. Cytology specimens (including fine needle aspirates) will not be accepted for CLDN18.2 examination. If archival tissue samples from several points of time are available, the most recent one is preferred. Patients with a lower expression level or with CLDN18.2-negative cancers are not eligible.

Trial part-specific inclusion criteria:

For Part 1A: Patients with solid tumors, for which there is no available standard therapy likely to confer clinical benefit, or the patient is not a candidate for such available therapy. Patients must have received all available standard therapies and failed at least first-line standard of care therapy prior to enrolment. Measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Eligible tumor types are gastric cancer, GEJ and esophageal adenocarcinoma, pancreatic, biliary tract (cholangiocarcinoma and gallbladder cancer), and mucinous ovarian cancers. Additionally, patients with specific tumors (including colorectal cancer, non small-cell lung cancer, gastric subtype of endocervical adenocarcinoma) where there is scientific evidence that the CLDN18.2 could be elevated can be tested for CLDN18.2 expression.

For Part 1B: Patients with advanced pancreatic adenocarcinoma or cholangiocarcinoma who are eligible for treatment with nab-paclitaxel and gemcitabine. Measurable or evaluable disease per RECIST 1.1.

Key exclusion criteria:

* Receiving: radiotherapy, chemotherapy, or molecularly-targeted agents within 3 weeks or 5 half-lives (whichever is longer) of the start of trial treatment; immunotherapy/monoclonal antibodies within 3 weeks of the start of trial treatment (excluding BNT141); nitrosoureas, antibody-drug conjugates, or radioactive isotopes within 6 weeks of the start of trial treatment. Palliative radiotherapy will be allowed.
* Receives concurrent systemic (oral or IV) steroid therapy >10 mg prednisone daily or its equivalent for an underlying condition. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is permitted.
* Major surgery within 4 weeks before the first dose of BNT141.
* Prior treatment with a CLDN18.2 targeting monoclonal antibodies (mAb) other than BNT141.
* Ongoing or active infection requiring IV treatment with anti-infective therapy that has been administered less than 2 weeks prior to the first dose of BNT141.
* Side effects of any prior therapy or procedures for any medical condition not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.5.0 Grade ≤ 1, with the exception of anorexia, fatigue, hyperthyroidism, hypothyroidism, and peripheral neuropathy, which must have recovered to ≤ Grade 2. Alopecia of any grade is allowed.
* Current evidence of new or growing brain or leptomeningeal metastases during screening. Patients with known brain or leptomeningeal metastases may be eligible if they have:

  * Radiotherapy, surgery or stereotactic surgery for the brain or leptomeningeal metastases.
  * No neurological symptoms (excluding Grade ≤ 2 neuropathy).
  * Stable brain or leptomeningeal disease on the computer tomography or magnet resonance imaging scan within 4 weeks before signing the informed consent form.
  * Not undergoing acute corticosteroid therapy or steroid taper.

Additional inclusion and exclusion criteria did apply (please refer to the clinical study protocol for detailed information).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (7):
- United States (4):
  - City of Hope, Duarte, California
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - START, San Antonio, Texas
- Canada (3):
  - University of Montreal - Centre Hospitalier de l´Université de Montréal, Montreal
  - St. Michaels Hospital, Toronto
  - Princess Margaret Cancer Centre - University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahr-Mahmud H, Ellinghaus U, Stadler CR, Fischer L, Lindemann C, Chaturvedi A, Diekmann J, Woll S, Biermann I, Hebich B, Scharf C, Siefke M, Roth AS, Rao M, Brettschneider K, Ewen EM, Sahin U, Tureci O. Preclinical characterization of an mRNA-encoded anti-Claudin 18.2 antibody. Oncoimmunology. 2023 Oct 16;12(1):2255041. doi: 10.1080/2162402X.2023.2255041. eCollection 2023. PMID 37860278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 patients (6 from Canada and 9 from the USA) were screened while 13 patients (5 patients and 8 patients respectively from two countries) were enrolled in this study and 2 patients failed screening (primary reason inclusion/exclusion criteria not met). All patients were enrolled into Part 1A of this study and received BNT141.
Pre-assignment Details: Adult patients with CLDN18.2-positive tumors. CLDN18.2 positivity was determined by a central laboratory during the pre-screening phase using a validated immunohistochemistry assay and was defined as moderate (50-75%)-to-strong (more than 75%) CLDN18.2 expression.
  No participant was enrolled in the planned Part 1B and Part 2 of this study.
Groups:
- BNT141 Monotherapy - 0.15 mg/kg: The number of patients from Part 1A treated with BNT141 0.15 mg/kg. BNT141 was administered IV as monotherapy once every three weeks.
- BNT141 Monotherapy - 0.30 mg/kg: The number of patients from Part 1A treated with BNT141 0.30 mg/kg. BNT141 was administered IV as monotherapy once every three weeks.
- BNT141 Monotherapy - 0.45 mg/kg: The number of patients from Part 1A treated with BNT141 0.45 mg/kg, corresponding to an intermediate dose level.
  BNT141 was administered IV as monotherapy once every three weeks.
- BNT141 Monotherapy - 0.60 mg/kg: The number of patients from Part 1A treated with BNT141 0.60 mg/kg. BNT141 was administered IV as monotherapy once every three weeks.
Period: Overall Study
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Started | 3 | 3 | 4 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 3
Not completed — Study termination by the sponsor | 0 | 1 | 2 | 2
Not completed — Death | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set - All patients who received investigational medicinal product (IMP) (i.e., at least one dose of BNT141)
Groups:
- Total: Total of all reporting groups
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2 | 0 | 4
  >=65 years | 1 | 3 | 2 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (15.52) | 73.7 (7.02) | 58.3 (11.35) | 74.0 (6.24) | 64.9 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 3
  Male | 2 | 2 | 3 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 3 | 4 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 2 | 2 | 5
  United States | 3 | 2 | 2 | 1 | 8
Eastern Cooperative Oncology Group performance score (ECOG PS) [Number; unit: Participants] — ECOG PS grading defined as follows:
  * Grade 0 - Fully active, able to carry on all pre-disease performance without restriction
  * Grade 1 - Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * Grade 2 - Ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50% of waking hours
  Participants
    ECOG PS 0 | 0 | 2 | 2 | 0 | 4
    ECOG PS 1 | 3 | 1 | 2 | 3 | 9
    ECOG PS 2 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is the patient's body weight in kilograms divided by the square of the patient's height in meters.
  kg/m^2 | 32.56 (7.120) | 24.41 (1.541) | 20.46 (4.888) | 24.67 (5.530) | 25.14 (6.42)
Number of prior systemic cancer therapies per patient [Mean (Standard Deviation); unit: number of therapies] | 3.7 (1.15) | 3.3 (2.52) | 3.8 (0.50) | 1.7 (0.58) | 3.2 (1.46)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Treatment-emergent Adverse Events (TEAEs) Within a Patient Including Grade ≥ 3, Serious, Fatal TEAE by Relationship
Description: All TEAEs are included, i.e., AEs with an onset date on or after the first dose of BNT141 (if the AE was absent before the first dose) or worsened after the first dose of BNT141 (if the AE was present before the first dose). AEs with an onset date >60 days after the last dose of BNT141 are included only if assessed as related to BNT141 by the investigator.
  Intensity of AEs was graded according to the NCI CTCAE v5.0, i.e.,:
  Grade 1 - Mild, Grade 2 - Moderate, Grade 3 - Severe, Grade 4 - Life-threatening consequences; urgent urgent intervention indicated, Grade 5 - Death related to AE
Time Frame: From start of BNT141 treatment until the second Safety Follow-up Visit (60 ± 7 days after last dose), up to 30 weeks.
Population: Safety Set - All patients who received investigational medicinal product (IMP) (i.e., at least one dose of BNT141)
Measure: Number; unit: participants
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3
participants
  Any TEAE | 3 | 3 | 4 | 3
  Related TEAE | 3 | 3 | 4 | 3
  Grade ≥3 TEAE | 0 | 2 | 2 | 1
  Related Grade ≥3 TEAE | 0 | 0 | 0 | 1
  Any serious TEAE | 1 | 1 | 1 | 2
  Related serious TEAE | 0 | 1 | 0 | 1
  TEAE of special interest | 0 | 1 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0

2. Primary Outcome: Occurrence of Dose Reductions and Discontinuation of BNT141 Due to TEAEs
Description: All TEAEs are included, i.e., AEs with an onset date on or after the first dose of BNT141 (if the AE was absent before the first dose) or worsened after the first dose of BNT141 (if the AE was present before the first dose). AEs with an onset date >60 days after the last dose of BNT141 are included only if assessed as related to BNT141 by the investigator
Time Frame: From start of BNT141 treatment until the second Safety Follow-up Visit (60 ± 7 days after last dose), up to 30 weeks.
Population: Safety Set - All patients who received investigational medicinal product (IMP) (i.e., at least one dose of BNT141)
Measure: Number; unit: participants
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3
participants
  TEAE leading to treatment discontinuation | 0 | 0 | 0 | 0
  Related TEAE leading to treatment discontinuation | 0 | 0 | 0 | 0
  TEAE leading to study drug interruption | 0 | 2 | 1 | 1
  Related TEAE leading to study drug interruption | 0 | 2 | 0 | 1
  TEAE leading to dose reduction | 0 | 0 | 0 | 0
  Related TEAE leading to dose reduction | 0 | 0 | 0 | 0
  TEAE leading to dose rate reduction | 0 | 0 | 0 | 0
  Related TEAE leading to dose rate reduction | 0 | 0 | 0 | 0

3. Primary Outcome: Occurrence of Dose-limiting Toxicities (DLTs) Within a Patient During the DLT Evaluation Period
Description: Serious AEs, non-serious Grade ≥ 3 non-hematological and hematological AEs as defined per DLT criteria and clinically significant abnormal laboratory values Grade ≥ 3 were collected and considered a DLT if assessed by the investigator to be at least possibly related to BNT141. Toxicities clearly not related to BNT141 (e.g., progressive disease, comorbidity, etc.) were not considered a DLT. The NCI CTCAE v.5.0 was used to grade the intensity of AEs.
Time Frame: First treatment cycle (From first dose up to 21 days after first dose)
Population: Safety Set - All patients who received investigational medicinal product (IMP) (i.e., at least one dose of BNT141)
Measure: Number; unit: participants
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3
participants | 0 | 0 | 0 | 0

4. Secondary Outcome: RiboMab PK Parameter - Area Under the Concentration Time Curve (AUC)
Description: Intact RiboMab (full-length and fully assembled antibody) PK serum samples were collected and analyzed.
  AUC (0-tau), AUC (0-inf) and AUC (0-504) were estimated from serum concentration data from Cycle 1 using non-compartmental analysis.
  AUC (0-inf): Area under the drug concentration-time curve, from time zero to infinity.
  AUC (0-504): Area under the drug concentration-time curve, from time zero to 504 hours after the start of the infusion.
  AUC (0-tau): Area under the drug concentration-time curve, from time zero over the dosing interval at steady-state (Tau = 504 hours corresponding to 3-weeks administration) after the start of the infusion.
Time Frame: First treatment cycle (From first dose up to 21 days after first dose)
Population: PK Set - All patients with baseline and at least one valid on-treatment/post-treatment PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3
h*ng/mL
  AUC (0-tau) | 1613407.9486 (50) | 5798293.4278 (30) | 5499389.8684 (40) | 5244472.7649 (60)
  AUC (0-inf): number analyzed (Participants) | 3 | 3 | 3 | 3
  AUC (0-inf) | 2166227.7262 (50) | 9838894.4371 (50) | 9128700.3987 (50) | 6739801.3745 (50)
  AUC (0-504): number analyzed (Participants) | 3 | 3 | 3 | 3
  AUC (0-504) | 1615489.8795 (50) | 5736526.2444 (30) | 6253473.9330 (40) | 5283854.6455 (60)

5. Secondary Outcome: RiboMab PK Parameter - Clearance
Description: Intact RiboMab (full-length and fully assembled antibody) PK serum samples were collected and analyzed.
  Clearance was estimated from serum concentration from Cycle 1 data using non-compartmental analysis.
Time Frame: First treatment cycle (From first dose up to 21 days after first dose)
Population: PK Set - All patients with baseline and at least one valid on-treatment/post-treatment PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
L/h | 0.0065 (60) | 0.0021 (40) | 0.0036 (50) | 0.0066 (70)

6. Secondary Outcome: RiboMab PK Parameter - Volume of Distribution at Steady State (Vss)
Description: Intact RiboMab (full-length and fully assembled antibody) PK serum samples were collected and analyzed.
  Volume of distribution at steady state (Vss) was estimated as mean residence time calculated using last measured concentration (MRT inf) * CL.
Time Frame: First treatment cycle (From first dose up to 21 days after first dose)
Population: PK Set - All patients with baseline and at least one valid on-treatment/post-treatment PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
L | 2.2103 (70) | 1.1099 (40) | 1.5656 (20) | 2.0340 (80)

7. Secondary Outcome: RiboMab PK Parameter - Maximum Serum Drug Concentration (Cmax)
Description: Intact RiboMab (full-length and fully assembled antibody) PK serum samples were collected and analyzed.
  Cmax was estimated from serum concentration from Cycle 1 data using non-compartmental analysis.
Time Frame: First treatment cycle (From first dose up to 21 days after first dose)
Population: PK Set - All patients with baseline and at least one valid on-treatment/post-treatment PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3
ng/mL | 5844.7265 (60) | 17829.5955 (40) | 24001.7233 (40) | 19801.0462 (60)

8. Secondary Outcome: RiboMab PK Parameter - Time to Reach Cmax (Tmax)
Description: Intact RiboMab (full-length and fully assembled antibody) PK serum samples were collected and analyzed.
  Tmax was estimated from serum concentration from Cycle 1 data using non-compartmental analysis.
Time Frame: First treatment cycle (From first dose up to 21 days after first dose)
Population: PK Set - All patients with baseline and at least one valid on-treatment/post-treatment PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3
hours | 59.80362 (20) | 61.02810 (20) | 68.18978 (30) | 54.72251 (20)

9. Secondary Outcome: RiboMab PK Parameter - Concentration at the End of a Dosing Interval (Taken Directly Before Next Administration) (Ctrough)
Description: Intact RiboMab (full-length and fully assembled antibody) PK serum samples were collected and analyzed.
  Ctrough was estimated from serum concentration from Cycle 1 data using non-compartmental analysis.
  Ctrough values are available for participants treated with dose level 1 and dose level 2 only.
Time Frame: Before start of Cycle 3 (plasma sample taken directly before BNT141 Cycle 3 administration)
Population: PK Set - All patients with baseline and at least one valid on-treatment/post-treatment PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg
Number analyzed (Participants) | 1 | 2
ng/mL | 3516.7500 (NA) — Only data from one participant was analyzed. | 3734.1225 (50)

10. Secondary Outcome: RiboMab PK Parameter - Half-time (t½)
Description: Intact RiboMab (full-length and fully assembled antibody) PK serum samples were collected and analyzed.
  T½ was estimated from serum concentration from Cycle 1 data using non-compartmental analysis.
Time Frame: First treatment cycle (From first dose up to 21 days after first dose)
Population: PK Set - All patients with baseline and at least one valid on-treatment/post-treatment PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
hours | 236.9571 (10) | 366.7979 (50) | 304.9024 (30) | 214.7214 (10)

11. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the number of patients in whom a complete response (CR) or partial response (PR), per RECIST 1.1 is confirmed as best overall response.
Time Frame: From start of first dose of BNT141 until end of trial or start of a new anti-cancer therapy, up to 30 weeks
Population: Data were not available for this endpoint due to early termination of the study meaning ORR could not be determined.
  Most participants were followed up for efficacy for a short period of time while on study (≤ 6 weeks), therefore there was insufficient follow-up for efficacy in most participants to conduct a meaningful assessment of ORR. As per statistical analysis plan, the analysis of secondary efficacy endpoint ORR was removed from the study analysis.
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the number of patients in whom a CR or PR or stable disease ([SD], per RECIST 1.1, SD assessed at least 6 weeks after first dose) is observed as best overall response.
Time Frame: From start of first dose of BNT141 until end of trial or start of a new anti-cancer therapy, up to 30 weeks
Population: Data were not available for this endpoint due to early termination of the study meaning DCR could not be determined.
  Most participants were followed up for efficacy for a short period of time while on study (≤ 6 weeks), therefore there was insufficient follow-up for efficacy in most participants to conduct a meaningful assessment of DCR. As per statistical analysis plan, the analysis of secondary efficacy endpoint DCR was removed from the study analysis.
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Duration of Response (DoR)
Description: DOR was defined as the time from first objective response (CR or PR per RECIST 1.1) to first occurrence of objective tumor progression (progressive disease per RECIST 1.1) or death from any cause, whichever occurs first.
Time Frame: From start of first dose of BNT141 until end of trial or start of a new anti-cancer therapy, up to 30 weeks
Population: Data were not available for this endpoint due to early termination of the study meaning DoR could not be determined.
  Most participants were followed up for efficacy for a short period of time while on study (≤ 6 weeks), therefore there was insufficient follow-up for efficacy in most participants to conduct a meaningful assessment of DoR. As per statistical analysis plan, the analysis of secondary efficacy endpoint DoR was removed from the study analysis.
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Deaths and SAEs: All events from the signing of the trial-specific informed consent from until the second Safety Follow-up Visit, up to 33 weeks. Other AEs: All TEAEs, i.e., AEs reported from the start of study drug treatment until the second Safety Follow-up Visit, up to 30 weeks.
Description: Other AEs: All TEAEs, i.e., AEs with an onset date on or after the first dose of BNT141 (if the AE was absent before the first dose) or worsened after the first dose of BNT141 (if the AE was present before the first dose). AEs with an onset date >60 days after the last dose of BNT141 are included only if assessed as related to BNT141 by the investigator.
Arm/Group | BNT141 Monotherapy - 0.15 mg/kg | BNT141 Monotherapy - 0.30 mg/kg | BNT141 Monotherapy - 0.45 mg/kg | BNT141 Monotherapy - 0.60 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 2/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/4 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT141 Monotherapy - 0.15 mg/kg (N=3) | BNT141 Monotherapy - 0.30 mg/kg (N=3) | BNT141 Monotherapy - 0.45 mg/kg (N=4) | BNT141 Monotherapy - 0.60 mg/kg (N=3)
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT141 Monotherapy - 0.15 mg/kg (N=3) | BNT141 Monotherapy - 0.30 mg/kg (N=3) | BNT141 Monotherapy - 0.45 mg/kg (N=4) | BNT141 Monotherapy - 0.60 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3 | 2
Chills (General disorders) | 1 | 2 | 2 | 1
Drug intolerance (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1
Cytokine release syndrome (Immune system disorders) | 3 | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

Principal Investigators respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT04683939/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT04683939/SAP_003.pdf